CLINICAL TRIAL: NCT06270862
Title: A Digital Active Aging Training Program for Older Adults
Acronym: AAT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Toronto Metropolitan University (Other)
Collaborators: Social Sciences and Humanities Research Council of Canada (Other); AGE-WELL and the Canadian Frailty Network (Unknown); Cogniciti (Unknown); Cognifit (Unknown); Aging in Cloud (Unknown)
Responsible Party: Principal Investigator, Lixia Yang, Professor, Toronto Metropolitan University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Health Services Research
Other Study IDs: SSHRC-PEG2023-AAT
Record Dates: First submitted 2024-01-01; First posted 2024-02-21 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Healthy Aging; Cognitive Change; Psychological Stress; Loneliness; Social Interaction
Keywords: Older adults; Active aging; Digital intervention; Resilience
MeSH Terms: conditions — Stress, Psychological | interventions — Cognitive Training; Exercise; Drug Interactions

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Active aging with resilience (AR) (Experimental): In the "active aging with resilience (AR)" condition, participants will complete physical, cognitive, and social engagement training modules, starting with a 15-min resilience-building module.
  Interventions: Behavioral: Resilience training; Behavioral: cognitive training; Behavioral: physical exercise; Behavioral: social interaction
- Active aging without resilience (AA) (Active Comparator): The traditional "active aging" (AA) training involves the same multi-domain active aging training without the initial resilience-building module, which will be replaced by watching 15 minutes of educational video on topics such as health, nature or travel.
  Interventions: Behavioral: cognitive training; Behavioral: physical exercise; Behavioral: social interaction
- Workshop training (WT) (Placebo Comparator): The "workshop training" (WT) control condition involves workshops following the same 4-week schedule on aging-related topics.
  Interventions: Behavioral: workshop series

INTERVENTIONS:
Behavioral: Resilience training — Receive mini course on what is resilience and how to use different exercises to be more resilient in life.
  Arms: Active aging with resilience (AR)
Behavioral: cognitive training — Play games that trains attention, memory and planning using the services provided by CogniFit.
  Arms: Active aging with resilience (AR); Active aging without resilience (AA)
Behavioral: physical exercise — Engage in age-appropriate physical exercises.
  Arms: Active aging with resilience (AR); Active aging without resilience (AA)
Behavioral: social interaction — Engage in social discussion with peers in the group.
  Arms: Active aging with resilience (AR); Active aging without resilience (AA)
Behavioral: workshop series — Watch a series of workshops targeting the older adult population.
  Arms: Workshop training (WT)

SUMMARY:
The proposed project aims to develop and validate a multi-dimensional digital active aging program integrated with resilience to promote the biopsychosocial functions of older adults aged 60, including Chinese older immigrants in Canada (Study 1) and English-speaking White Canadian older adults (Study 2).

The proposed study takes a typical pretest-training-posttest design. Pretest and posttest: a battery of outcome measures on physical, psychological, and social functions will be administered to all participants. Data will also be used to identify sociodemographic risk predictors for outcome variables (i.e., biopsychosocial functions and resilience). Training: the participants will be randomly assigned to three arms to receive 4 weeks of 16 training/practice/control treatment sessions delivered via Zoom.

In the "active aging with resilience (AR)" condition, participants will complete physical, cognitive, and social engagement training modules, starting with a 30-min resilience-building module. The traditional "active aging" (AA) training involves the same multi-domain active aging training without the initial resilience-building module. The "workshop training" (WT) control condition involves workshops following the same 4-week schedule on aging-related topics.

DETAILED DESCRIPTION:
Objectives:

1. to develop a multi-domain digital active aging training program through Zoom to promote active aging; and
2. to evaluate whether adding a resilience-building module would enhance the active aging training efficacy to mitigate the lingering detrimental impacts of the pandemic

Sample:

For Study 1, the investigators will recruit 120 Mandarin-speaking healthy older Chinese immigrants (aged 60+, Chinese migrants) through WeChat(a popular instant messaging app among Chinese)/email/lab website social media channels (e.g., Facebook, Twitter) from the community partners (see a list attached). For Study 2, we will recruit 120 English-speaking healthy White Canadian older adults (aged 60+) through TMSPSS (the senior participant pool at Toronto Metropolitan University) or advertisements.

Overall Design and Procedure:

Informed consent will be collected. The proposed study will take a traditional pretest-intervention-posttest design including three phases of research activities. In Phase 1 (pretest), the investigators will administer a large battery of outcome measures including physical, psychological (emotional and cognitive), and social function measures to assess the baseline performance. The data collected at pretest also addresses the first sub-objective to identify sociodemographic risk predictors for the biopsychosocial functions and resilience among Chinese older immigrants in Canada. In Phase 2 (intervention), participants will be randomly assigned to an "active aging with resilience", an "active aging", and a "workshop" control condition. They will go through 4 weeks of 8 sessions of training/control treatment delivered virtually through Zoom/YouTube and 8 sessions of offline self-practice. In Phase 3 (posttest), all participants who completed the intervention programs will complete the same battery of the outcome measures as administered at the pretest session. Their performance on the outcome measures at posttest will be compared against pretest to evaluate the efficacy of the training programs.

Intervention:

The virtually-delivered intervention program will be developed based on previous studies and practices that proved to be effective in resilience-building and active.

During the 4-week training period delivered through Zoom/YouTube, participants in the "active aging with resilience" group will complete 8 sessions (approximately 1.5 hours per session and 2 sessions per week) of active aging training program integrated with a resilience-building module. Each session will start with a 15-min session of resilience building activities modified from positive psychology resilience-building activities that promotes various resilience characters (e.g., gratitude, forgiveness, grit etc.). This will be followed by the 1-hour multi-dimensional active aging training activities, including progressive "aging in motion" physical and nutrition training (e.g., age-appropriate "Choose to move" physical workout on-line videos), cognitive training with executive function and speed based on a customized module on CogniFit website, socialization and social engagement (e.g., discussion on the topic and session, followed by homework on volunteering, calling friends/families, community activity participation etc.), and combined bio-psycho-social multi-component training (e.g., performing a cognitive tasks such as counting backwards or memorizing names while doing physical exercise in a virtual socialization setting). Participants in the "active aging" group will receive the same training except that the initial 15-min resilience-building activities will be replaced by warmup activities such as watching some pre-selected video on active aging and completing a quiz afterwards. Both the "active aging with resilience" and traditional "active aging" group will also engage in 8 offline practice sessions where they follow instructions to practice and repeat the last completed modules. Finally, participants in the receptive "workshop" control group will attend 8 virtual workshops or watching workshop videos (following the same 4-week schedule as the two training groups) on different aging-related topics such as physical health, mental health, cognitive wellbeing, emotional regulation, social engagement, and resilience. Each workshop will take approximately 1.5 hours (including 30 min for questions). They will also review and watch the replays of last workshops and take a short survey question after each review session. All these activities will be delivered virtually via Zoom/YouTube in groups of 10-15 individuals.

Data Analysis Plan To identify active aging and resilience predictors, a set of explorative multivariate linear regression models will be conducted on the data collected at the pretest session, with all sociodemographic as predictors and outcome measure performance as dependent variables. To evaluate the relative efficacy of the active aging intervention programs, a 3 (condition) by 2 (session) mixed model analysis of variances (ANOVA) models will be conducted on each outcome variable, after controlling for potential sociodemographic covariates. For comparison and clarity purposes, if the outcome measures within each function domain demonstrates similar patterns, the investigators will calculate a composite outcome variable based on the z-scores of all involved measures to index the performance level of that specific functional domain. This composite score will be used as the outcome variable in the ANOVA. In light of the literature, the investigators hypothesized that the "active aging with resilience" training will produce larger and wider benefits relative to the "active aging" training, both compared against the receptive "workshop" control condition.

ELIGIBILITY:
Inclusion Criteria:

Study 1(Chinese group):

1. Aged 65 or over and healthy
2. Chinese migrant (e.g., Canadian citizens, immigrants, visitors that are born and raised in the Chinese culture)
3. Can speak, read and write Mandarin
4. Having access to a computer that has internet and allows Zoom meeting attendance

Study 2(Canadian group):

1. Aged 65 or over and healthy
2. White Canadian citizen
3. Can speak, read and write English
4. Having access to a computer that has internet and allows Zoom meeting attendance

Exclusion Criteria:

1. Scored 10 or above on the Short blessed test (SBT)
2. Unfit for light physical exercises
3. Without access to a computer and internet
4. With current or previous mental health diagnosis

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2024-04-08 (Actual); Primary Completion 2024-10-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Exercise Self-efficacy level (ESES) | (1) pre-test (2) through study completion, an average of 1 month (3) 1-month post study completion
  (out of 40) higher score means better self-efficacy at carrying out regular physical activities and exercise.
the 5-item World Health Organization WellBeing Index (WHO-5) | (1) pre-test (2) through study completion, an average of 1 month (3) 1-month post study completion
  (out of 25) higher score indicates better overall self-perception of wellbeing in the past 2 weeks
Kessler Psychological Distress Scale (K10) | (1) pre-test (2) through study completion, an average of 1 month (3) 1-month post study completion
  (out of 50) higher score indicates worse overall mental health
Multidimensional Scale of Perceived Social Support (MSPSS) | (1) pre-test (2) through study completion, an average of 1 month (3) 1-month post study completion
  (out of 7) higher score indicates higher levels of self-precepted social support
Conner-Davidson Resilience Scale 10-item (CD RISC-10) | (1) pre-test (2) through study completion, an average of 1 month (3) 1-month post study completion
  (out of 40) higher score indicates higher resilience in face of difficulty in life.
Emotional regulation Questionnaire (ERQ) | (1) pre-test (2) through study completion, an average of 1 month (3) 1-month post study completion
  Cognitive reappraisal (out of 42) and expressive suppression (out of 28). Higher score indicates higher inclination to use this facet to control their emotions.
Positive and Negative Affect Schedule (PANAS) | (1) pre-test (2) through study completion, an average of 1 month (3) 1-month post study completion
  Positive affect (out of 50) and negative affect (out of 50). Higher score indicates feelings of higher levels of the positive/negative affect at the moment.
Visual working memory test | (1) pre-test (2) through study completion, an average of 1 month (3) 1-month post study completion
  Assessed using computerized games from CogniFit. Higher score indicates better visual short-term memory and memory span.
Divided attention test | (1) pre-test (2) through study completion, an average of 1 month (3) 1-month post study completion
  Assessed using computerized games from CogniFit. Higher score indicates better ability to divide attention between two competing tasks.
Visual memory test | (1) pre-test (2) through study completion, an average of 1 month (3) 1-month post study completion
  Assessed using computerized games from CogniFit. Higher score indicates better ability to memorize and recognize shapes and sequence order of visual object.
Stroop test | (1) pre-test (2) through study completion, an average of 1 month (3) 1-month post study completion
  Assessed using computerized games from CogniFit. Higher score indicates better ability to inhibit irrelevant information in tasks.
Sustained attention to response test | (1) pre-test (2) through study completion, an average of 1 month (3) 1-month post study completion
  Assessed using computerized games from CogniFit. Higher score indicates better ability to sustain attention to show rapid response to targets when present.

SECONDARY OUTCOMES:
Satisfaction with life scale (SWLS) | (1) pre-test (2) through study completion, an average of 1 month (3) 1-month post study completion
  (out of 35) higher score indicates higher self-perception of life satisfaction
Instrumental Activities of Daily Living(IADL) | (1) pre-test (2) through study completion, an average of 1 month (3) 1-month post study completion
  (out of 8) higher score indicates better ability to carry out daily physical activity
The 6-item De Jong Gierveld Loneliness Scale | (1) pre-test (2) through study completion, an average of 1 month (3) 1-month post study completion
  (out of 30) higher score indicates higher levels of loneliness
The Brief Approach/Avoidance Coping Questionnaire (BACQ) | (1) pre-test (2) through study completion, an average of 1 month (3) 1-month post study completion
  approach (out of 30) and avoidance (out of 30) scores. Higher score in each category indicates their inclination to act in relation to problems and illness.

CONTACTS AND LOCATIONS:
Overall Officials: Lixia Yang, PhD, Principal Investigator — Toronto Metropolitan University
Locations (1):
- Cognitive Aging Lab, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Armitage R, Nellums LB. COVID-19 and the consequences of isolating the elderly. Lancet Public Health. 2020 May;5(5):e256. doi: 10.1016/S2468-2667(20)30061-X. Epub 2020 Mar 20. No abstract available. PMID 32199471
- [Background] Carstensen LL, Shavit YZ, Barnes JT. Age Advantages in Emotional Experience Persist Even Under Threat From the COVID-19 Pandemic. Psychol Sci. 2020 Nov;31(11):1374-1385. doi: 10.1177/0956797620967261. Epub 2020 Oct 26. PMID 33104409
- [Background] Bandura, A. (2006). Guide for constructing self-efficacy scales. In: Urdan T, Pajares F (eds.) Self-Efficacy Beliefs of Adolescents. New York, NY, USA: Information Age Publishing.
- [Background] Chappell, N. L. & Havens, B. (1980). Old and Female: Testing the Double Jeopardy Hypothesis. The Sociological Quarterly, 21(2), 157-171,
- [Background] Diener E, Emmons RA, Larsen RJ, Griffin S. The Satisfaction With Life Scale. J Pers Assess. 1985 Feb;49(1):71-5. doi: 10.1207/s15327752jpa4901_13. PMID 16367493
- [Background] Dong X. Elder abuse in Chinese populations: a global review. J Elder Abuse Negl. 2015;27(3):196-232. doi: 10.1080/08946566.2015.1039154. Epub 2015 Apr 15. PMID 25874889
- [Background] Finset, A., Steine, S., Haugli, L., Steen, E., Laerum, E. (2002). The brief approach/avoidance coping questionnaire: Development and validation. Psychology, health & medicine, 7(1):75-85
- [Background] Galea S, Merchant RM, Lurie N. The Mental Health Consequences of COVID-19 and Physical Distancing: The Need for Prevention and Early Intervention. JAMA Intern Med. 2020 Jun 1;180(6):817-818. doi: 10.1001/jamainternmed.2020.1562. No abstract available. PMID 32275292
- [Background] Gao, Z. (2021). Unsettled Belongings: Chinese immigrants' mental health nulnerability as a symptom of international politics in the COVID-19 pandemic. Journal of Humanistic Psychology, 61(2), 198-218. https://doi.org/10.1177/0022167820980620
- [Background] De Jong Gierveld, J., & Van Tilburg, T. (2006). A 6-Item Scale for Overall, Emotional, and Social Loneliness: Confirmatory Tests on Survey Data. Research on Aging, 28(5), 582-598. https://doi.org/10.1177/0164027506289723
- [Background] Kanning, M., Schlicht, W. (2008). A bio-psycho-social model of successful aging as shown through the variable "physical activity". European Review of Aging and Physical Activity, 5, 79-87. https://doi.org/10.1007/s11556-008-0035-4
- [Background] Kessler RC, Andrews G, Colpe LJ, Hiripi E, Mroczek DK, Normand SL, Walters EE, Zaslavsky AM. Short screening scales to monitor population prevalences and trends in non-specific psychological distress. Psychol Med. 2002 Aug;32(6):959-76. doi: 10.1017/s0033291702006074. PMID 12214795
- [Background] Lai DW, Surood S. Chinese health beliefs of older Chinese in Canada. J Aging Health. 2009 Feb;21(1):38-62. doi: 10.1177/0898264308328636. PMID 19144968
- [Background] Lai, D. W. L., Daoust G., Li, L. (2014). Understanding elder abuse and neglect in aging Chinese immigrants in Canada. The Journal of Adult Protection, 16(5):322-34. DOI:10.1108/JAP-03-2014-0006
- [Background] Lawton MP, Brody EM. Assessment of older people: self-maintaining and instrumental activities of daily living. Gerontologist. 1969 Autumn;9(3):179-86. No abstract available. PMID 5349366
- [Background] Lovibond PF, Lovibond SH. The structure of negative emotional states: comparison of the Depression Anxiety Stress Scales (DASS) with the Beck Depression and Anxiety Inventories. Behav Res Ther. 1995 Mar;33(3):335-43. doi: 10.1016/0005-7967(94)00075-u. PMID 7726811
- [Background] Mendoza-Ruvalcaba NM, Arias-Merino ED. "I am active": effects of a program to promote active aging. Clin Interv Aging. 2015 May 5;10:829-37. doi: 10.2147/CIA.S79511. eCollection 2015. PMID 26005337
- [Background] Na L, Yang L, Mezo PG, Liu R. Age disparities in mental health during the COVID19 pandemic: The roles of resilience and coping. Soc Sci Med. 2022 Jul;305:115031. doi: 10.1016/j.socscimed.2022.115031. Epub 2022 May 13. PMID 35649300
- [Background] Perez-Rojo G, Lopez J, Noriega C, Velasco C, Carretero I, Lopez-Frutos P, Galarraga L. A multidimensional approach to the resilience in older adults despite COVID-19. BMC Geriatr. 2022 Oct 11;22(1):793. doi: 10.1186/s12877-022-03472-y. PMID 36221056
- [Background] Qian M, Wu Q, Wu P, Hou Z, Liang Y, Cowling BJ, Yu H. Anxiety levels, precautionary behaviours and public perceptions during the early phase of the COVID-19 outbreak in China: a population-based cross-sectional survey. BMJ Open. 2020 Oct 8;10(10):e040910. doi: 10.1136/bmjopen-2020-040910. PMID 33033099
- [Background] Qiu J, Shen B, Zhao M, Wang Z, Xie B, Xu Y. A nationwide survey of psychological distress among Chinese people in the COVID-19 epidemic: implications and policy recommendations. Gen Psychiatr. 2020 Mar 6;33(2):e100213. doi: 10.1136/gpsych-2020-100213. eCollection 2020. PMID 32215365
- [Background] Roussey, K. (2018). Why these university students love living with seniors. CBC. Published September 6, 2018. Accessed May 8, 2020. https://www.cbc.ca/news/health/student-senior-university-mcmaster-housing-co-generational-1.4811115
- [Background] Rowe JW, Kahn RL. Human aging: usual and successful. Science. 1987 Jul 10;237(4811):143-9. doi: 10.1126/science.3299702.
- [Background] Singelis' T. M. (1994). The measurement of independent and interdependent self-construals. Personality and Social Psychology Bulletin' 20' 580-591.
- [Background] Smith BW, Dalen J, Wiggins K, Tooley E, Christopher P, Bernard J. The brief resilience scale: assessing the ability to bounce back. Int J Behav Med. 2008;15(3):194-200. doi: 10.1080/10705500802222972. PMID 18696313
- [Background] Su C, Yang L, Dong L, Zhang W. The Psychological Well-Being of Older Chinese Immigrants in Canada amidst COVID-19: The Role of Loneliness, Social Support, and Acculturation. Int J Environ Res Public Health. 2022 Jul 15;19(14):8612. doi: 10.3390/ijerph19148612. PMID 35886464
- [Background] United Nations (2013). Department of Economic and Social Affairs, Population Division. World Population Ageing 2013. New York, NY, USA: United Nations.
- [Background] Wu B. Social isolation and loneliness among older adults in the context of COVID-19: a global challenge. Glob Health Res Policy. 2020 Jun 5;5:27. doi: 10.1186/s41256-020-00154-3. eCollection 2020. PMID 32514427
- [Background] Yang L. Practice-oriented retest learning as the basic form of cognitive plasticity of the aging brain. J Aging Res. 2011;2011:407074. doi: 10.4061/2011/407074. Epub 2011 Oct 31. PMID 22132328
- [Background] Yang L. Maintained and Delayed Benefits of Executive Function Training and Low-Intensity Aerobic Exercise Over a 3.5-Year Period in Older Adults. Front Aging Neurosci. 2022 Jul 1;14:905886. doi: 10.3389/fnagi.2022.905886. eCollection 2022. PMID 35847677
- [Background] Yang L, Gallant SN, Wilkins LK, Dyson B. Cognitive and Psychosocial Outcomes of Self-Guided Executive Function Training and Low-Intensity Aerobic Exercise in Healthy Older Adults. Front Aging Neurosci. 2020 Nov 19;12:576744. doi: 10.3389/fnagi.2020.576744. eCollection 2020. PMID 33328958
- [Background] Yang L, Kandasamy K, Na L, Zhang W, Wang P. Perceived and Experienced Anti-Chinese Discrimination and Its Associated Psychological Impacts Among Chinese Canadians During the Wave 2 of the COVID-19 Pandemic. Psychol Health Med. 2024 Jan-Jun;29(1):108-125. doi: 10.1080/13548506.2022.2142947. Epub 2022 Nov 6. PMID 36336783
- [Background] Yang L, Yu L, Kandasamy K, Wang Y, Shi F, Zhang W, Wang PP. Non-Pathological Psychological Distress among Mainland Chinese in Canada and Its Sociodemographic Risk Factors amidst the Pandemic. Healthcare (Basel). 2022 Nov 21;10(11):2326. doi: 10.3390/healthcare10112326. PMID 36421650
- [Background] Yin J, Lassale C, Steptoe A, Cadar D. Exploring the bidirectional associations between loneliness and cognitive functioning over 10 years: the English longitudinal study of ageing. Int J Epidemiol. 2019 Dec 1;48(6):1937-1948. doi: 10.1093/ije/dyz085. PMID 31056641
- [Background] Zhang W. Perceptions of elder abuse and neglect by older Chinese immigrants in Canada. J Elder Abuse Negl. 2019 Aug-Dec;31(4-5):340-362. doi: 10.1080/08946566.2019.1652718. Epub 2019 Aug 8. PMID 31394984
- [Background] Zimet, G. D., Dahlem, N. W., Zimet, S. G., Farley, G. K. (1988). The Multidimensional Scale of Perceived Social Support. Journal of Personality Assessment, 52(1), 30-41. https://doi.org/10.1207/s15327752jpa5201_2
- See also: Choose to Move at Home video modules — https://vimeo.com/user101392358
- See also: 23 resilience building activities & exercises for adults. Resilience & Coping, Positive Psychology — https://positivepsychology.com/resilience-activities-exercises